CLINICAL TRIAL: NCT04649723
Title: A Single-Center, Single-Arm, Open-Label, Fixed-Sequence Phase I Drug-Drug Interaction Clinical Study of the Effect of Rifampicin on Pharmacokinetics of SHR1459 in Chinese Healthy Subjects.
Brief Title: Drug-Drug Interaction of SHR1459 With a Strong CYP3A Index Inducer (Rifampicin)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SHR1459-I-105
Record Dates: First submitted 2020-11-10; First posted 2020-12-02 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2020-11

CONDITIONS: Healthy Subjects, Drug-drug Interaction, Pharmacokinetics, SHR1459
MeSH Terms: interventions — Rifampin

STUDY DESIGN:
Intervention Model Description: To observe the effect of rifampicin on the pharmacokinetics of SHR1459 and to evaluate the safety of SHR1459, rifampicin and their coadministration in Chinese healthy subjects. The subjects will take SHR1459 at first single dose, then washout period, and take it at second single dose after multiple administration of rifampicin to get a full induction condition.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rifampicin 600 mg + SHR1459 Tablets 200 mg (Experimental)
  Interventions: Drug: Rifampin; Drug: SHR1459
- SHR1459 tablets 200 mg (Active Comparator)
  Interventions: Drug: SHR1459

INTERVENTIONS:
Drug: Rifampin — single oral dose, 600 mg, fasted.
  Arms: Rifampicin 600 mg + SHR1459 Tablets 200 mg
Drug: SHR1459 — single oral dose, 200 mg, fasted.

SUMMARY:
This drug-drug interaction (DDI) study had been designed to investigate the effect of a strong CYP 3A index fan-inducer rifampicin on the pharmacokinetics of SHR1459 in Chinese healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent before the trial, and fully understand the trial content, process and possible adverse reactions;
2. Ability to complete the study as required by the protocol;
3. Healthy male or female subjects aged 18 to 45 (including 18 and 45) at the date of signing the informed consent;
4. Body weight ≥50 kg for male and≥ 45 kg for female, and body mass index (BMI) within the range of 19 ~ 26 kg /m2 (including 19 and 26);
5. In females, documented surgical sterilization, postmenopausal status for at least 1 year (follicle stimulating hormone [FSH] > 40 mIU/mL serum at Screening), or agreement to use an approved form of contraception
6. In males, agreement to avoid sperm donation for 3 months days after the dose of SHR1459
7. Liver function test results must be below the upper limit of normal.
8. Participants must agree to refrain from donation of whole blood and other blood products from 90 days prior to screening.
9. Heart rate ≥60 bpm.
10. GFR≥90 mL/min/1.73m2.

Exclusion Criteria:

1. Loss of more than 400 mL blood during the 3 months before the trial (eg, as a blood donor)
2. Allergic constitution;
3. History of drug use, or drug abuse screening positive;
4. Alcoholic or often drinkers;
5. A smoker with 5 cigarettes per day for more than 90 days;
6. Positive serology for hepatitis B surface antigen (HBsAg) and HCV (healthy participants), anti-treponema pallidum virus (TP), or antihuman immunodeficiency virus (HIV) Type 1 and Type 2 (all subjects)
7. Use of any drugs or substances known to be inhibitors or inducers of CYP3A within 90 days from the first dose or 5 half-lives, if known, of the drugs or substances, whichever is greater, prior to SHR1459 administration and during the study.
8. A clear medical history of important primary organ diseases such as nervous system, cardiovascular system, urinary system, digestive system, respiratory system, metabolism and musculoskeletal system.
9. Abnormal clinical laboratory tests and clinical significance judged by the investigator or other clinical findings showing the following diseases, including but not limited to gastrointestinal tract, kidney, liver, nerve, blood, endocrine, tumor, lung, immune, mental or cardiovascular and cerebrovascular diseases.
10. Use of grapefruit or marmalade in 2 weeks prior to admission to the clinical unit, as reported by the subject.
11. Major surgery within 6 months before screening.
12. Woman in breastfeeding and pregnancy and with egg donation plan, and man with sperm donation plan in 6 months after follow-up in the trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) for SHR1459. | predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24h for Day1 and Day9
Area Under the Plasma Concentration-time Curve from 0 to any time before the last quantifiable concentration (AUC0-t) for SHR1459. | predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24h for Day1 and Day9
Area Under the Plasma Concentration-time Curve from 0 to infinite time (AUCinf) for SHR1459. | predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24h for Day1 and Day9

SECONDARY OUTCOMES:
Other pharmacokinetics parameters of SHR1459: Tmax, T1/2, CL, Vd, etc | predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24h for Day1 and Day9
The incidence and severity of adverse events/serious adverse events (based on NCI-CTCAE 5.0): Laboratory indicators, 12-lead electrocardiogram (ECG), physical examination, vital signs, etc. | Baseline up to 14 days post last dose, up to approximately 2 month

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu HengRui Medicine Co., Ltd., Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No